CLINICAL TRIAL: NCT04906837
Title: Pre TAVI Membranous Septum Measurement Predicts High Grade Iatrioventricular Conduction Disorders in Patients With Specific Pacemaker Implanted After TAVI. The STIM TAVI-MS Study
Acronym: STIM TAVI MS
Status: Completed | Type: Observational
Sponsor: Association de Recherche en Cardiologie des Alpes (Other)
Responsible Party: Sponsor
Other Study IDs: AlpinARC
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Conduction Disturbance; Trans Aortic Valve Implantation (TAVI)
Keywords: membranous septum; valve implantation height; predictive factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Trans aortic valve implantation — Measurement of the membranous septum on the pre TAVI scanner and the valve implantation height

SUMMARY:
Conduction disturbances are a major complication of TAVI. There is no predictor of post-TAVI conduction disorder. The study of the membranous septum on the pre-TAVI scanner and the valve implantation height are promising and little studied data on the occurrence of post-TAVI conduction disorders.

DETAILED DESCRIPTION:
After being developed for the treatment of aortic stenosis in inoperable patients, trans aortic valve implantation (TAVI) techniques and devices have gradually improved, and its use can now be considered in low-risk populations. . However, the need for pacemaker implantation after TAVI remains one of the most common complications, and this issue needs to be addressed before further expanding the TAVI indications.

Implantation of PM after TAVI is associated with increased morbidity and mortality, and there are no formal predictors of these conduction disturbances. Some studies suggest that the existence of preoperative conduction disturbances (eg, right bundle branch block or 1st degree AVB) are associated with greater PM implantation or greater reliance on ventricular pacing.

Other studies have focused on anatomical measurements such as the height of the membranous septum obtained on the pre TAVI scanner, calcifications of the aortic ring and the depth of the valve implantation obtained on the angiography of the TAVI procedure. . The depth of valve implantation in relation to the height of the membranous septum would be a predictor of conduction disorders and PM implantation post TAVI.

Anatomically, the left branch of the bundle of HIS originates approximately 6 mm below the aortic annulus. Implantation of TAVI can affect the conduction tissues and lead to conduction abnormalities where the penetrating portion of the HIS emerges on the surface of the LV flushing chamber. The farther away the emerging part of the HIS is from the ring, the less likely it is that an implant will encroach on it, and impair conduction.

Because the emerging part of the bundle of His is "sandwiched" between the membranous septum and the posterior crest of the muscular septum, the lower end of the membranous septum provides an anatomical landmark for the left ventricular exit point of the bundle of His, with the length of the membranous septum equivalent to the distance aortic ring - bundle of HIS.

The STIM TAVI study showed that 30% of patients implanted with a post-TAVI pacemaker did not have high-grade AVB beyond 7 days post-implantation. Patients with early AVB (D1-D7) were at high risk of developing late AVB. The study did not identify a population at low risk of late-onset AVB, nor any pre-TAVI clinical or paraclinical criteria predictive of post-TAVI AVB.

The study of the anatomy of the membranous septum and the height of implantation of the aortic prosthesis in the STIM TAVI population would make it possible to analyze new predictive criteria for late AVB (after D7).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Patients included in the STIM TAVI study with full follow-up (not excluded from STIM TAVI for lack of data)
* Patients who did not object to the use of CT and angiography data

Exclusion Criteria:

* Oral opposition to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients included in the STIM TAVI study with full follow-up (not excluded from STIM TAVI for lack of data)
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
One late high-grade AVB | between day 7 to one year
  Presence of at least one late high-grade AVB episode

SECONDARY OUTCOMES:
CT and angiographic measurements, | one year
  Feasibility of CT and angiographic measurements,
intra and inter observer variability | one year
  intra and inter observer variability.

CONTACTS AND LOCATIONS:
Locations (1):
- CH Annecy Genevois, Annecy, France

IPD SHARING:
Plan to Share IPD: Undecided